CLINICAL TRIAL: NCT01500603
Title: Prospective, Randomized, Multicentric, Comparative Trial of Two Devices in Surgical Treatment of Post-radical Prostatectomy Stress Urinary Incontinence: Periurethral Pro-ACTTM Balloons and AdvanceXP(TM) Retrourethral Male Sling
Brief Title: Periurethral Pro-ACTTM Balloons vs Retrourethral AdvanceXP(TM) Male Sling for Post-prostatectomy Incontinence
Acronym: BALLANCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion in the study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P100143
Record Dates: First submitted 2011-12-23; First posted 2011-12-28 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Stress Urinary Incontinence
Keywords: post-radical prostatectomy; stress urinary incontinence; periurethral Pro-ACT balloons; AdvanceXP retrourethral male sling
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Patients will receive AdvanceXP retrourethral male sling implantation under general or loco-regional anaesthesia, by perineal approach. The sling is placed via transobturator route
  Interventions: Device: AdvanceXP Male sling device
- Active comparator (Active Comparator): Patients will receive Pro-ACT balloons implantation under general or loco-regional anaesthesia, by perineal approach. The balloons are placed under X-ray control laterally to the urethra, under the bladder neck. The extremity of the device (titanium port), linked to the balloon, is located subcutaneously in the scrotum. During post-operative visits, readjustments of the volume of the balloons will be made under local anaesthesia. The volume will be increased or decreased according to the patients symptoms.
  Interventions: Device: Pro-ACT balloon device

INTERVENTIONS:
Device: AdvanceXP Male sling device — Patients will receive AdvanceXP retrourethral male sling (polypropylene mesh) implantation under general or loco-regional anaesthesia, by perineal approach. The sling is placed via transobturator route.
  Arms: Experimental
Device: Pro-ACT balloon device — Patients will receive Pro-ACT balloons implantation under general or loco-regional anaesthesia, by perineal approach. The balloons are placed under X-ray control laterally to the urethra, under the bladder neck. The extremity of the device (titanium port), linked to the balloon, is located subcutaneously in the scrotum. During post-operative visits, readjustments of the volume of the balloons will be made under local anaesthesia. The volume will be increased or decreased according to the patients symptoms.
  Arms: Active comparator

SUMMARY:
Background: Periurethral Pro-ACT balloons and retrourethral AdvanceXP(TM) male sling have been presented as efficient treatments for management of stress urinary incontinence (SUI) following radical prostatectomy (RP), but no comparative study of these two techniques has been published. The investigators aims were to compare the efficacy of the two devices and provide data about their cost effectiveness.

Hypothesis: The study is based on the superiority hypothesis that AdvanceXP male slings is more efficacious than Pro-ACT balloons at one year follow-up.

Primary objective: The primary objective of this study is to compare the efficacy of the AdvanceXP retrourethral male sling and periurethral Pro-ACT balloons management of SUI after RP at one year follow-up.

Secondary objectives:

* Comprehensive comparative medical evaluation of the two devices in terms of efficacy
* Complete evaluation of the side effects of the two techniques
* Evaluation of the quality of life
* Evaluation of patient satisfaction
* Cost-effectiveness study of the device (total cost over one year of each of the two techniques, differential cost-effectiveness ratio (cost adjusted by QALY), differential cost-effectiveness ratio in terms adjusted to success rate, recommendations that can be made for assessing the potential coverage by the French healthcare system) Population: Patients with history of RP without cancer recurrence, presenting pure SUI on urodynamics (without detrusor overactivity), of mild to moderate degree (24hour pad-test < 300g).

Study design: This is a prospective, randomized, multicentric (9 tertiary reference centers), comparative trial of the two devices (with a superiority hypothesis). The total number of subjects required is 240 and inclusion period is 12 months. Follow-up consists in 4 visits at 1, 3, 6 and 12 months, with data collection (pad use, uroflowmetry, quality of life validated questionnaires ICIQ-SF and EQ-5D, 24-hr pad test, patient satisfaction with PGI-I and report of any secondary effect). Statistical evaluation is carried out at the end of the follow-up, in intent to treat.

Medical evaluation:

Main criterion:failure of the treatment, defined by reduction of less than 50% of incontinence on 24-hr pad test, explantation of the device or implantation of a new surgical device for SUI.

Secondary outcome criteria

* pad usage per day
* quantitative reduction of the 24hr-pad test
* complications (infection, erosion, hematoma, acute urinary retention)
* number of re-interventions or re-admissions during follow-up
* quality of life measured by the ICIQ-SF questionnaire
* patient satisfaction by the PGI-I questionnaire

Economic evaluation:

* Study of the total cost over one year in each case
* Adjustment of cost of each device to quality of life (QALY evaluation)
* Cost effectiveness study
* Proposals will be made to state at which level the two devices should be covered by the healthcare system.

DETAILED DESCRIPTION:
Background: Stress urinary incontinence (SUI) is a common adverse event of radical prostatectomy (RP) for localized prostate cancer and can dramatically impact quality of life. Management of SUI after RP is based on conservative measures and pelvic floor muscle training. In case of failure of this first line therapy, surgical treatment is required. In recent years, periurethral Pro-ACT balloons and retrourethral AdvanceXP male sling have been proven to be efficient to manage SUI after RP in case of mild to moderate symptoms. Pro-ACT balloons are placed under general anesthesia via a perineal approach, laterally to the membranous urethra under the bladder neck. This device results in an external compression of the urethra. Further adjustment of the compression is possible under local anesthesia since the balloons are linked to a subcutaneous titanium port. AdvanceXP male sling is placed under general anesthesia via a perineal approach, by transobturator route, and results in a suspension of the membranous urethra relocating the bladder neck. If multiple reports have claimed for the efficacy of these two devices, they have never been compared in a prospective comparative trial. Our aims were to compare the efficacy of the two devices and provide data about their cost effectiveness.

Hypothesis: The study is based on the superiority hypothesis that Advance male slings is more efficacious than Pro-ACT balloons at one year follow-up.

Objectives:

The primary objective of this study is to compare the efficacy of the Advance retrourethral male sling and periurethral Pro-ACT balloons for post-prostatectomy stress urinary incontinence (SUI) management.

The secondary objectives of this work are:

* Comprehensive medical evaluation of these two emerging devices in terms of efficiency using the usual criteria in the field of urinary incontinence
* Complete evaluation of the side effects of the two techniques
* Evaluation of the quality of life
* Cost-effectiveness study of the device (Total cost over one year of each of the two techniques, differential cost-effectiveness ratio (cost adjusted by QALY), differential cost-effectiveness ratio in terms adjusted to success rate, recommendations that can be made for assessing the potential coverage by the French healthcare system

Population: The study concerns patients presenting SUI following radical prostatectomy for prostate cancer. Patients must be older than 18, without cancer recurrence, and must present pure SUI on urodynamics (without detrusor overactivity), and mild to moderate incontinence (24hour pad-test < 300g). Every patient showing urethral stricture at preoperative cystoscopy is excluded from the study.

Study design: This is a prospective, randomized, multicentric (9 tertiary reference centers), comparative trial of the two devices (with a superiority hypothesis). The study begins with a 12 months inclusion period. The total number of subjects required is 240. At the end of the inclusion process, a randomization in two arms is carried out. Follow-up consists in 4 visits at 1, 3, 6 and 12 months, with data collection (pad use, uroflowmetry, quality of life validated questionnaires ICIQ-SF and EQ-5D, 24-hr pad test, patient satisfaction with PGI-I and report of any secondary effect). Statistical evaluation is carried out at the end of the follow-up, in intent to treat.

Medical evaluation:

The main criterion of the study is failure of the treatment, defined by reduction of less than 50% of incontinence on 24-hr pad test, explantation of the device or implantation of a new surgical device for SUI management in the year after operation.

Secondary criteria are focused on efficacy and tolerance and evaluated during follow-up at 1, 3, 6 and 12 months on the following criteria:

* pad usage per day
* quantitative reduction of the 24hr-pad test
* complications (infection, erosion, hematoma, acute urinary retention)
* number of re-interventions or re-admissions during follow-up
* quality of life measured by the ICIQ-SF questionnaire
* patient satisfaction by the PGI-I questionnaire The statistical evaluation on the main criterion will be carried out by the chi-square test. Variables with a known predictive value on efficiency (radiation therapy, severity of incontinence) will be studied by logistic regression then multivariate analysis. The results will be adjusted on the centers (multicentric study). The quantitative variables will be compared by Mann-Whitney test.

Economic evaluation: The economic evaluation will be carried out according to the following manner:

* A study of the total cost over one year of each device, based on the data collected during the clinical trial and including all the events that required medical care (visits, complications, reinterventions, readmissions), but also the cost of pads (not supported by healthcare system, and only supported by the patient).
* From this study led on cost and of the collection of quality of life data, the cost of each device will be adjusted to quality of life (QALY evaluation)
* A cost effectiveness study will also be lead, by adjusting cost to success rate of each technique
* Proposals will be made to state at which level the two devices should be covered by the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient presenting mild to moderate stress urinary incontinence (20g < 72 hours pad-test < 300g) following radical prostatectomy more than 1 year ago.
* Patient capable of roaming, independent and capable of using toilet without any trouble.
* Patients able to answer to questionnaire and communicate in French
* Informed consent
* Patients with social security

Exclusion Criteria:

* Uncontrolled prostatic adenocarcinoma or PSA > 1 ng/ml
* Maximum urinary flow rate < 15 ml/sec
* Postvoid residual volume > 150 ml
* Urinated volume in 24h > 3000 ml
* Uninhibited detrusor contractions associated with leakage during the preoperative urodynamic assessment (realized under anticholinergic if the patient is usually under this medication)
* Severe incontinence (Pad test > 300g/24h)
* History of artificial urinary sphincter
* Known neurologic bladder dysfunction
* History of neurological disease which can interfere with the urinary symptoms
* Presence of a urethral stenosis or of an anastomotic stricture during the preoperative endoscopy.
* Previous treatment with pelvic radiation therapy in 6 months before inclusion
* Uncontrolled urinary tract infection
* Patients affected by an infiltrative bladder tumour
* Patients with bladder stones
* Severe constitutional hemorrhagic disease or haemophilia
* Deep depression of immune system
* Severe renal impairment or obstructive pathology of the upper urinary tract with severe renal impairment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
failure of the treatment, defined by reduction of less than 50% of incontinence on 24-hr pad test, explantation of the device or implantation of a new surgical device for SUI management in the year after operation | 12 months after surgical treatment

SECONDARY OUTCOMES:
complications | 1, 3 6 and 12 months after surgical treatment
  * pad usage per day
  * quantitative reduction of the 24hr-pad test
  * complications (infection, erosion, hematoma, acute urinary retention)
  * number of re-interventions or re-admissions during follow-up
  * quality of life measured by the ICIQ-SF questionnaire
  * patient satisfaction by the PGI-I questionnaire
Cost-effectiveness study of the device | 12 months after surgical treatment
  [Total cost over one year of each of the two techniques, differential cost-effectiveness ratio (cost adjusted by QALY), differential cost-effectiveness ratio in terms adjusted to success rate, recommendations that can be made for assessing the potential coverage by the French healthcare system]

CONTACTS AND LOCATIONS:
Overall Officials: François Haab, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service d'urologie, Hôpital Tenon, Paris, France